CLINICAL TRIAL: NCT02847832
Title: Prospective Validation and Comparison of Subjective Assessment, the International Ovarian Tumor Analysis (IOTA) ADNEX Model, Logistic Regression Model LR2, Simple Rules and the Risk of Malignancy Index (RMI) for Discrimination Between Benign and Malignant Adnexal Masses in the Hands of Ultrasound Examiners With Different Levels of Experience
Brief Title: Prospective Validation and Comparison of Different Ultrasound Methods for Discrimination Between Benign and Malignant Ovarian/Tubal Masses Prior to Surgery
Acronym: IOTA7
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Dirk Timmerman, Prof. Dr., KU Leuven
Other Study IDs: IOTA7 s59207
Record Dates: First submitted 2016-07-15; First posted 2016-07-28 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Patients With Adnexal Mass Prior to Surgery
Keywords: Adnexal Diseases; Ovary; Ovarian Neoplasms; Ovarian Cysts; Ovarian Diseases; Ultrasonography; Ultrasonography, Doppler; Diagnosis; Early Diagnosis; Early Detection of Cancer; Genital Neoplasms, Female; Genital Diseases, Female; Urogenital Neoplasms; Cysts; Endocrine System Diseases; Gonadal Disorders; Neoplasms; Endocrine Gland Neoplasms; International Ovarian Tumor Analysis; Simple Rules; Preoperative evaluation; Prediction Models; Logistic Regression Models; Mathematical Models; Adnexal Masses; Ovarian Tumors; Risk of Malignancy
MeSH Terms: conditions — Adnexal Diseases; Ovarian Neoplasms; Ovarian Cysts; Ovarian Diseases; Disease; Genital Neoplasms, Female; Genital Diseases, Female; Urogenital Neoplasms; Cysts; Endocrine System Diseases; Gonadal Disorders; Neoplasms; Endocrine Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for CA-125 measurement
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Standardized transvaginal ultrasound examination

SUMMARY:
The ability of different methods to discriminate between benign and malignant adnexal masses has been compared in a meta-analysis showing that the IOTA Simple Rules and the IOTA logistic regression model LR2 were superior to RMI and to all other methods for predicting malignancy in an adnexal mass included in the meta-analysis. However, a fair comparison of methods requires them to be applied on the same tumor population.

The general objective of this study is to prospectively validate the Simple Rules, ADNEX, the Simple Rules risk model, LR2, and RMI on a large multicenter dataset to allow direct comparison of these tools.

IOTA7 is an international multicenter prospective observational study including different types of ultrasound centers and examiners with different levels of ultrasound experience. In total, about 1700 adnexal masses with histological outcome will be included in IOTA 7.

DETAILED DESCRIPTION:
Ovarian cancer is a common and lethal disease for which early detection and treatment in high volume centers and by specialized clinicians is known to improve survival. Hence, accurate methods to preoperatively characterize the nature of an ovarian tumor are pivotal.

The best ultrasound method for discrimination between benign and malignant adnexal masses is subjective assessment, i.e. subjective evaluation of ultrasound findings. Subjective assessment, however, requires a very experienced ultrasound examiner. More objective methods may be preferred by less experienced examiners who are not confident with using subjective assessment. The Risk of Malignancy Index (RMI) is one such method. There are also more recently developed methods. The International Ovarian Tumor Analysis (IOTA) group have created logistic regression models (LR1, LR2, and the ADNEX model) including clinical and ultrasound information to calculate the likelihood of malignancy in adnexal masses.

The IOTA group has also suggested simple ultrasound rules that can be used to classify adnexal masses as benign or malignant.

The ability of different methods to discriminate between benign and malignant adnexal masses has been compared in a meta-analysis showing that the IOTA Simple Rules and the IOTA logistic regression model LR2 were superior to RMI and to all other methods for predicting malignancy in an adnexal mass included in the meta-analysis. However, a fair comparison of methods requires them to be applied on the same tumor population.

The general objective of this study is to prospectively validate the Simple Rules, ADNEX, the Simple Rules risk model, LR2, and RMI on a large multicenter dataset to allow direct comparison of these tools. The patients will be examined by operators of varying levels of experience, such that the investigators can study how experience might affect diagnostic performance.

IOTA7 is an international multicenter prospective observational study including different types of ultrasound centers and examiners with different levels of ultrasound experience. In total, about 1700 adnexal masses with histological outcome will be included in IOTA 7.

Patients with a known or suspected adnexal mass examined with transvaginal (or transrectal if vaginal is not possible) ultrasound by an IOTA certified ultrasound examiner and confirmed to have an adnexal mass judged not to be physiological but likely to undergo surgery (primarily planned for surgical management based on subjective assessment by the ultrasound investigator) will be recruited consecutively Upon inclusion in the study, an oral or written (depending on the requirements of the local Ethics Committee) informed consent is obtained from the patient.

Data collection is done through the web-based clinical data miner (CDM) software. Data are stored on a secure server.

First, clinical information about the patient is entered into CDM. Second, the ultrasound examiner provides a diagnosis based on subjective assessment, and notes the suggested management. Third, detailed ultrasound information needed for the different models to be validated is entered. When these data have been frozen (so they can no longer be changed) the examiner gets access to the results of the Simple Rules and ADNEX. The ultrasound examiner then records whether these results make him/her change the management suggested on the basis of subjective assessment. If so the new management is specified.

Gold standard for validation of discriminative ability and calibration is the histology of the adnexal mass within 180 days after the ultrasound examination following surgical removal by laparotomy or laparoscopy as considered appropriate by the surgeon. In case of malignancy, the stage of the malignant tumors using the classification of the International Federation of Gynecology and Obstetrics (FIGO) is noted.

ELIGIBILITY:
Inclusion Criteria:

* Any woman presenting with an adnexal mass judged not to be physiological and likely to undergo surgery (primarily planned for surgical management based on subjective assessment by the ultrasound examiner; however, the ultrasound examiner is allowed to change the advised management to conservative management after the results of Simple Rules or ADNEX are known).
* Pregnant patients can be included but will be analysed separately.
* Patients finally selected for conservative management can be included but will not be used for all statistical analyses.
* For patients selected for surgery, delay of surgery is not an exclusion criterion for this study, but for selected objectives only those patients in whom surgery was performed within 180 days after the ultrasound examination will be assessed.
* Patients can be selected at any age, but for patients <18 years old, a guardian's permission should be obtained.
* Patients that only underwent transabdominal scanning can be included in the study, but will be analysed separately.

Exclusion Criteria:

* Previous bilateral adnexectomy
* Denial or withdrawal of informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a known or suspected adnexal mass examined with transvaginal (or transrectal if vaginal is not possible) ultrasound by an IOTA certified ultrasound examiner and confirmed to have an adnexal mass judged not to be physiological but likely to undergo surgery (primarily planned for surgical management based on subjective assessment by the ultrasound investigator).
  Different types of ultrasound centers (general gynecologic outpatient clinic or specialized ultrasound centers) and examiners with different levels of ultrasound experience will be involved.
Sampling Method: Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative likelihood ratios with regard to detection of malignancy for different ultrasound methods | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
AUCs for discrimination between benign and malignant masses for prediction models. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.

SECONDARY OUTCOMES:
Flexible calibration curves based on local regression (loess) to assess calibration of the estimated risks on malignancy given by the risk prediction models. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Sensitivity, specificity, positive and negative likelihood ratios with regard to detection of malignancy for different ultrasound methods, in hands of examiners with different level of experience. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
AUCs for prediction models, in hands of examiners with different level of experience. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Sensitivity, specificity, positive and negative likelihood ratios with regard to detection of malignancy for different ultrasound methods, where the Simple Rules are inconclusive. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
AUCs for prediction models, where the Simple Rules are inconclusive. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Change of the suggested management based on subjective assessment depending on the level of expertise of the ultrasound examiner, after results of the Simple Rules have been shown. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Polytomous discrimination index for the ADNEX model to discriminate between different classes of histology. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
AUCs for each pair of outcome categories using the conditional risk method for the ADNEX model to discriminate between different classes of histology. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Multinomial calibration curves for the ADNEX model to predict benign tumors, borderline tumors, stage 1 primary ovarian cancer, stage 2-4 primary ovarian cancer and metastatic cancer. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Adjusted odds ratios with regard to malignancy for selected ultrasound characteristics, mainly papillation characteristics, in the subgroup of unilocular cysts with papillations. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
Sensitivity and specificity with regard to malignancy at different risk cutoffs, for a risk prediction model in unilocular cysts with papillations based on a limited number of variables selected a priori. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.
AUC for a risk prediction model in unilocular cysts with papillations based on a limited number of variables selected a priori. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 180 days after ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bourne, MD, PhD, Study Chair — Queen Charlotte's & Chelsea Hospital, Imperial College London, London, UNITED KINGDOM; Ben Van Calster, MSc, PhD, Study Chair — Department Development & Regeneration, KU Leuven, Leuven, BELGIUM; Ignace Vergote, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospitals KU Leuven, Leuven, BELGIUM; Lil Valentin, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, Skåne University Hospital, Malmö, SWEDEN; Antonia C Testa, MD, PhD, Study Chair — Unità Operativa di Ginecologia Oncologica Dipartimento Tutela della Salute della Donna e della Vita Nascente, Università Cattolica di Sacro Cuore, Roma, ITALY; Sabine Van Huffel, MSc, PhD, Study Chair — Department of electrical engineering (ESAT SCD-SISTA), KU Leuven, Heverlee-Leuven, BELGIUM
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Woo YL, Kyrgiou M, Bryant A, Everett T, Dickinson HO. Centralisation of services for gynaecological cancers - a Cochrane systematic review. Gynecol Oncol. 2012 Aug;126(2):286-90. doi: 10.1016/j.ygyno.2012.04.012. Epub 2012 Apr 13. PMID 22507534
- [Background] Engelen MJ, Kos HE, Willemse PH, Aalders JG, de Vries EG, Schaapveld M, Otter R, van der Zee AG. Surgery by consultant gynecologic oncologists improves survival in patients with ovarian carcinoma. Cancer. 2006 Feb 1;106(3):589-98. doi: 10.1002/cncr.21616. PMID 16369985
- [Background] Earle CC, Schrag D, Neville BA, Yabroff KR, Topor M, Fahey A, Trimble EL, Bodurka DC, Bristow RE, Carney M, Warren JL. Effect of surgeon specialty on processes of care and outcomes for ovarian cancer patients. J Natl Cancer Inst. 2006 Feb 1;98(3):172-80. doi: 10.1093/jnci/djj019. PMID 16449677
- [Background] Vernooij F, Heintz AP, Witteveen PO, van der Heiden-van der Loo M, Coebergh JW, van der Graaf Y. Specialized care and survival of ovarian cancer patients in The Netherlands: nationwide cohort study. J Natl Cancer Inst. 2008 Mar 19;100(6):399-406. doi: 10.1093/jnci/djn033. Epub 2008 Mar 11. PMID 18334710
- [Background] Valentin L, Hagen B, Tingulstad S, Eik-Nes S. Comparison of 'pattern recognition' and logistic regression models for discrimination between benign and malignant pelvic masses: a prospective cross validation. Ultrasound Obstet Gynecol. 2001 Oct;18(4):357-65. doi: 10.1046/j.0960-7692.2001.00500.x. PMID 11778996
- [Background] Timmerman D. The use of mathematical models to evaluate pelvic masses; can they beat an expert operator? Best Pract Res Clin Obstet Gynaecol. 2004 Feb;18(1):91-104. doi: 10.1016/j.bpobgyn.2003.09.009. PMID 15123060
- [Background] Jacobs I, Oram D, Fairbanks J, Turner J, Frost C, Grudzinskas JG. A risk of malignancy index incorporating CA 125, ultrasound and menopausal status for the accurate preoperative diagnosis of ovarian cancer. Br J Obstet Gynaecol. 1990 Oct;97(10):922-9. doi: 10.1111/j.1471-0528.1990.tb02448.x. PMID 2223684
- [Background] Kaijser J, Sayasneh A, Van Hoorde K, Ghaem-Maghami S, Bourne T, Timmerman D, Van Calster B. Presurgical diagnosis of adnexal tumours using mathematical models and scoring systems: a systematic review and meta-analysis. Hum Reprod Update. 2014 May-Jun;20(3):449-62. doi: 10.1093/humupd/dmt059. Epub 2013 Dec 9. PMID 24327552
- [Background] Timmerman D, Testa AC, Bourne T, Ferrazzi E, Ameye L, Konstantinovic ML, Van Calster B, Collins WP, Vergote I, Van Huffel S, Valentin L; International Ovarian Tumor Analysis Group. Logistic regression model to distinguish between the benign and malignant adnexal mass before surgery: a multicenter study by the International Ovarian Tumor Analysis Group. J Clin Oncol. 2005 Dec 1;23(34):8794-801. doi: 10.1200/JCO.2005.01.7632. PMID 16314639
- [Background] Van Calster B, Van Hoorde K, Valentin L, Testa AC, Fischerova D, Van Holsbeke C, Savelli L, Franchi D, Epstein E, Kaijser J, Van Belle V, Czekierdowski A, Guerriero S, Fruscio R, Lanzani C, Scala F, Bourne T, Timmerman D; International Ovarian Tumour Analysis Group. Evaluating the risk of ovarian cancer before surgery using the ADNEX model to differentiate between benign, borderline, early and advanced stage invasive, and secondary metastatic tumours: prospective multicentre diagnostic study. BMJ. 2014 Oct 15;349:g5920. doi: 10.1136/bmj.g5920. PMID 25320247
- [Background] Timmerman D, Testa AC, Bourne T, Ameye L, Jurkovic D, Van Holsbeke C, Paladini D, Van Calster B, Vergote I, Van Huffel S, Valentin L. Simple ultrasound-based rules for the diagnosis of ovarian cancer. Ultrasound Obstet Gynecol. 2008 Jun;31(6):681-90. doi: 10.1002/uog.5365. PMID 18504770
- [Background] Timmerman D, Van Calster B, Testa A, Savelli L, Fischerova D, Froyman W, Wynants L, Van Holsbeke C, Epstein E, Franchi D, Kaijser J, Czekierdowski A, Guerriero S, Fruscio R, Leone FPG, Rossi A, Landolfo C, Vergote I, Bourne T, Valentin L. Predicting the risk of malignancy in adnexal masses based on the Simple Rules from the International Ovarian Tumor Analysis group. Am J Obstet Gynecol. 2016 Apr;214(4):424-437. doi: 10.1016/j.ajog.2016.01.007. Epub 2016 Jan 19. PMID 26800772
- [Background] Installe AJ, Van den Bosch T, De Moor B, Timmerman D. Clinical data miner: an electronic case report form system with integrated data preprocessing and machine-learning libraries supporting clinical diagnostic model research. JMIR Med Inform. 2014 Oct 20;2(2):e28. doi: 10.2196/medinform.3251. PMID 25600863
- [Background] Heintz AP, Odicino F, Maisonneuve P, Quinn MA, Benedet JL, Creasman WT, Ngan HY, Pecorelli S, Beller U. Carcinoma of the ovary. FIGO 26th Annual Report on the Results of Treatment in Gynecological Cancer. Int J Gynaecol Obstet. 2006 Nov;95 Suppl 1:S161-92. doi: 10.1016/S0020-7292(06)60033-7. No abstract available. PMID 17161157
- [Derived] Landolfo C, Ceusters J, Valentin L, Froyman W, Van Gorp T, Heremans R, Baert T, Wouters R, Vankerckhoven A, Van Rompuy AS, Billen J, Moro F, Mascilini F, Neumann A, Van Holsbeke C, Chiappa V, Bourne T, Fischerova D, Testa A, Coosemans A, Timmerman D, Van Calster B. Comparison of the ADNEX and ROMA risk prediction models for the diagnosis of ovarian cancer: a multicentre external validation in patients who underwent surgery. Br J Cancer. 2024 Apr;130(6):934-940. doi: 10.1038/s41416-024-02578-x. Epub 2024 Jan 19. PMID 38243011